CLINICAL TRIAL: NCT01118507
Title: Trisomy of Chromosome 21 Diagnosis by High Output Sequencing of Foetal Circulating DNA in Mother Blood at First Trimester of Pregnancy.
Brief Title: Trisomy of Chromosome 21 Diagnosis by High Output Sequencing
Acronym: SEQ21
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 09071; 2009-A00908-49 (Registry Identifier: IDRCB)
Record Dates: First submitted 2010-04-28; First posted 2010-05-06 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Trisomy 21 - Translocation
Keywords: Trisomy of chromosome 21 diagnosis; first trimester of pregnancy; maternal blood; High output shotgun sequencing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fetal DNA in maternal blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TRISOMY: mothers of a trisomic fetus 21
- NORMAL KARYOTYPE: mothers of DISOMIQUE foetus 21

SUMMARY:
Demonstrate that the High output shotgun sequencing of the foetal DNA in the maternal blood could allow a complete discrimination between the mothers of a trisomic fetus 21 or a DISOMIQUE foetus 21 from the first quarter of the pregnancy, and so to obtain a reliable alternative in invasive procedure.

DETAILED DESCRIPTION:
Justification of the research :

The trisomy 21 is the most frequent cause of handicap of genetic origin with an incidence of 1.3/1 000 births which increases with the maternal age. Several strategies of antenatal screening were developed. The High Authority of Health recently recommended to propose to the pregnant women a 1st trimester combined screening, realized between 11+0 and 13+6 weeks of amenorrhoea, associating measure of the NUCALE translucency and dosage in maternal serum : PAPP-A (Pregnancy Associated Plasma Protein A) and βhCG (free β human Chorionic 1st trimester Gonadotrophin). However, the sensibility of these screening tests is about 80 % for 5 % of positive false. The diagnosis of aneuploidy is then established on a population classified at high risk, by a foetal karyotype (requiring an invasive procedure : biopsy of trophoblast or amniocentesis). A positive screening increase maternal and medical anxiety. Furthermore, the inappropriate combination of the tests is at the origin of numerous useless invasive procedures (national rate of amniocentesis of 11 %), at risk of foetal losses (0,5 in 1 %). This inflation of invasive procedures leads to so many losses of not affected children as trisomic children and to a badly known maternal morbidity.

Several studies showed that 10 % of the free DNA found from the first quarter of the pregnancy in the maternal plasma is of foetal origin and that this DNA is specific of the foetal nuclear DNA of the current pregnancy. This opened the way of a possible not invasive antenatal diagnosis of the foetal aneuploidy which collided during the last 10 years with the performances limited by the isolation and by the sequencing of the foetal DNA in the maternal plasma. A new technique of analysis by broadband sequencing of the DNA circulating in the maternal blood for the diagnosis of the most frequent aneuploid the trisomy 21 of which was brought back(reported). The High-output shotgun sequencing of all the DNA circulating in the maternal blood, then the reading and the identification of all the chromosome sequences allows to analyze the quantity of DNA resulting from the supernumerary chromosome, without necessity of differentiating maternal and foetal DNA. On the basis of very recent works 10, this excess of sequences resulting specifically from the chromosome 21 foetal supernumerary allows a discrimination completes between trisomy 21 and disomy 21. However, this study analyzed only 9 cases of trisomy 21 and the sampling of maternal blood were realized after the amniocentesis or the choriocenteses, what could artificially have increased the quantity of circulating foetal DNA.

Objectives :

Demonstrate that the High output shotgun sequencing of the foetal DNA in the maternal blood could allow a complete discrimination between the mothers of a trisomic fetus 21 or a DISOMIQUE fetus 21 from the first quarter of the pregnancy, and so to obtain a reliable alternative in invasive procedure.

Method Two public centres of antenatal screening were established to answer specifically the recommendations of the High Authority of Health and have the capacity to make 20 000 acts of screenings a year. All the women presenting a high risk (> 1/250) of aneuploidy and the candidates to an invasive procedure, will see suggesting participating in the study. The included patients will have a maternal blood sample before the invasive test. This taking will be put in on hold in-80°C after centrifugation following the recommended protocol. At the end of inclusion, the technic of analysis of the circulating DNA will be realized then blind by the laboratory on all the diagnosed cases (by usual invasive examination, or at the conclusion of the pregnancy) of trisomy 21 and on control representative of all the spectre of the levels of risk. A study of reproducibility of the quantification of the DNA of the chromosome 21 will be realized.

Number of subjects:

we plan to include 75 cases of trisomy 21 and 150 control cases with normal karyotype, what allows to detect a 99,9 % sensibility and a 99,99 % specificity with a power of at least 95 %.

Duration of the study:

these objectives are practicable in two years on the basis of the number of invasive takings realized in both center and an already realized study

Ethical Aspects: research on data and biological collection. No individual medical decision will be taken according to the estimated test.

Perspectives:

this new technique, if it is generalizable, would allow to limit the number of procedures of invasive diagnosis (amniocentesis and choriocentesis) which contain a significant risk of grave maternal and fetal complications, while optimizing the capacities of this screening.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* patient coming from one of multidisciplinary prenatal diagnosis center
* having à high risk of trisomy of chromosome 21 estimated by combine screening > 1/250
* 11 weeks of gestation or high
* accepting invasive prenatal diagnosis of chromosomal abnormalities
* accepting genetic analysis of blood circulating DNA
* Patient accepting to sign the enlightened assent

Exclusion Criteria:

* Patient of less than 18 years
* combine risk < 1/250
* refusing invasive prenatal diagnosis of chromosomal abnormalities
* refusing genetic analysis of blood circulating DNA
* Patient refusing to sign the enlightened assent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PREGNANT WOMEN
Sampling Method: Non-Probability Sample
Enrollment: 976 (Actual)
Dates: Start 2010-03; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The diagnostic performances of the quantification of the DNA resulting from the chromosome 21 by High output shotgun sequencing | 24 MONTHS
  The diagnostic performances(sensibility and specificity)of the quantification of the DNA resulting from the chromosome 21 by High-througput shotgun sequencing will be estimated in comparison with the results of the traditional cytogenetics obtained by culture of amniocytes or trophoblaste (gold standards).

SECONDARY OUTCOMES:
The time necessary for the treatments of samples: | 24 MONTHS
  this one will be estimated at the time means necessities to treat ten first ones and the last ten takings of the study
The cost by taking. | 24 MONTHS
  The cost in euro of the high output shotgun sequencing for one blood sample
The repeatability of the quantification: | 24 MONTHS
  this will be made by the realization of a double quantification, blind at ten drawn lots patients (these patients will be taken by two tubes instead of the only one and the laboratory will treat both tubes blind, as if they corresponded to two different patients.).

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT SALOMON, MCU PH, Principal Investigator — APHP
Locations (2):
- France (2):
  - Necker Enfants Malades, Paris
  - Chi Poissy St Germain, Poissy

REFERENCES:
- [Result] Alberti A, Salomon LJ, Le Lorc'h M, Couloux A, Bussieres L, Goupil S, Malan V, Pelletier E, Hyon C, Vialard F, Rozenberg P, Bouhanna P, Oury JF, Schmitz T, Romana S, Weissenbach J, Vekemans M, Ville Y. Non-invasive prenatal testing for trisomy 21 based on analysis of cell-free fetal DNA circulating in the maternal plasma. Prenat Diagn. 2015 May;35(5):471-6. doi: 10.1002/pd.4561. PMID 25643828